CLINICAL TRIAL: NCT03550781
Title: Does Inactive Takayasu Arteritis(NIH Criteria) Need Anti-inflammatory Treatment？
Brief Title: Anti-inflammatory Treatment for Inactive Takayasu Arteritis
Acronym: ATITA
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Xiongjing Jiang, Professor, Chinese Academy of Medical Sciences, Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-992
Record Dates: First submitted 2018-05-05; First posted 2018-06-08 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-06

CONDITIONS: Takayasu Arteritis; Anti-Inflammatory Agents
Keywords: Takayasu Arteritis; Anti-Inflammatory Agents; Positron Emission Tomography Computed Tomography
MeSH Terms: conditions — Takayasu Arteritis | interventions — Prednisone; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anti-inflammatory treatment group (Experimental): Prednisone and/or cyclophosphamide
  Interventions: Drug: Prednisone, cyclophosphamide
- Control group (No Intervention): No intervention

INTERVENTIONS:
Drug: Prednisone, cyclophosphamide — Prednisone 0.5mg/(kg•d) and/or cyclophosphamide 2mg/kg
  Arms: Anti-inflammatory treatment group

SUMMARY:
Currently, the traditional disease activity of Takayasu arteritis is mainly based on National Institutes of Health criteria and the inactive cases don't need anti-inflammatory treatment. However, pathologic findings showed that there was still inflammatory activity in the affected vessels, and the follow-up data also found significant lesion progression in some inactive cases. Sixty inactive Takayasu arteritis patients will be recruited to determine whether these individuals are active by screening new inflammatory markers in this study. New inflammatory markers included tumor necrosis factor,interleukin-2,interleukin-6,interleukin-8,interleukin-10,high-sensitivity C-reactive protein, and 18f-FDG positron emission tomograph. According to new inflammatory markers, sixty patients will be divided into two categories: inactive patients (n=20) and active patients (n=40). And then, Forty active patients diagnosed by new inflammatory markers will be randomly assigned to either anti-inflammatory therapy group or control group. The changes of inflammatory activity and lesion progression will be observed during one-year follow up in all 60 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Takayasu arteritis diagnosed by the American College of Rheumatology 1990 criteria;
2. Inactive Takayasu arteritis according to National Institutes of Health criteria;
3. Age ≥ 14 and ≤ 40 years old at the time of informed consent;
4. Patients or guardian agree to participate in the study.

Exclusion Criteria:

1. Active Takayasu arteritis according to National Institutes of Health criteria;
2. Poor compliance, intolerance to or poor response to hormone therapy;
3. Allergy to contrast agent;
4. Renal insufficiency (serum creatinine >133μmol/L), cardiac insufficiency (NYHA functional class III and IV) or abnormal liver function (Alanine transaminase >1.5 times upper limit of normal)

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-06-01 (Estimated); Primary Completion 2020-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Lesion progression | baseline and 12 months
  Progression of previous lesion degree>20% or new lesion

SECONDARY OUTCOMES:
Lesion progression | baseline, 3 months, 6 months, 9 months
  Progression of previous lesion degree>20% or new lesion
Changes in plasma concentration of tumor necrosis factor | baseline, 3 months, 6 months, 9 months and 12 months
Changes in plasma concentration of interleukin-2 | baseline, 3 months, 6 months, 9 months and 12 months
Changes in plasma concentration of interleukin-6 | baseline, 3 months, 6 months, 9 months and 12 months
Changes in plasma concentration of interleukin-8 | baseline, 3 months, 6 months, 9 months and 12 months
Changes in plasma concentration of interleukin-10 | baseline, 3 months, 6 months, 9 months and 12 months
Changes in plasma concentration of high-sensitivity C-reactive protein | baseline, 3 months, 6 months, 9 months and 12 months
Changes in 18F-fluorodeoxyglucose uptake by positron emission tomograph | baseline, 3 months, 6 months, 9 months and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiongjing Jiang, MD, Principal Investigator — Fuwai Hospital, National Center for Cardiovascular Disease, Chinese Academy of Medical Sciences and Peking Union Medical College

IPD SHARING:
Plan to Share IPD: Undecided